CLINICAL TRIAL: NCT06387147
Title: ORal Antibiotics in Acute Mesenteric Ischemia: a Multicenter Randomized Controlled Trial
Brief Title: ORal Antibiotics in Acute Mesenteric Ischemia
Acronym: ORIAMI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220818
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Acute Mesenteric Ischemia
Keywords: necrosis
MeSH Terms: conditions — Necrosis | interventions — Gentamicins; Metronidazole

STUDY DESIGN:
Intervention Model Description: double-blind Gentamicin + Metronidazole versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gentamicin + Metronidazole (Experimental): Gentamicin 80 mg Metronidazole 500mg 3 times per day during 14 days oral route or nasogastric tube or jejunostomy tube (in the case of an ostomy)
  Interventions: Drug: Gentamicin; Drug: Metronidazole
- Placebo (Placebo Comparator): Gentamicin placebo (2ml sodium chloride diluted 1/10 in a syringe of 20mL Metronidazole placebo in tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gentamicin — Gentamicin 80 mg 3 times per day during 14 days oral route or nasogastric tube or jejunostomy tube (in the case of an ostomy)
  Arms: Gentamicin + Metronidazole
Drug: Placebo — Gentamicin placebo (2ml sodium chloride diluted 1/10 in a syringe of 20mL Metronidazole placebo in tablets
  Arms: Placebo
Drug: Metronidazole — Métronidazole 500mg 3 times per day during 14 days oral route or nasogastric tube or jejunostomy tube (in the case of an ostomy)
  Arms: Gentamicin + Metronidazole

SUMMARY:
Acute mesenteric ischemia (AMI) is a life-threatening condition with an increasing incidence (7-13/100000 PY). The mortality of AMI is associated with the development and extent of transmural intestinal necrosis (IN), ranging from 25% without IN to 75% with IN. Given its potential reversibility, preventing the progression of AMI towards IN is now considered a primary therapeutic goal. Early management of AMI can thus avoid fatal outcomes and prevent lifelong complications such as short bowel syndrome. Following the results of a pilot study showing an improvement in survival and lower resection rates, our team created a first-of-its-kind intestinal stroke center (SURVI unit, Beaujon Hospital, Clichy, France) that provides 24/7 standardized multimodal and multidisciplinary care to AMI patients referred from all hospitals in the Paris region. As no randomized clinical trial has ever been conducted, the treatment offered by SURVI is based on pathophysiological knowledge and observational clinical data. AMI naturally progresses to sepsis, surgical complications, and multi-organ failure, direct consequences of IN. Features of sepsis are reported in up to 90% of AMI patients compared with 3-22% of patients with brain or myocardial ischemia, supporting a specific septic component in AMI. Experimental studies demonstrated reduced translocation and mortality in germ-free animals or after administration of oral antibiotics targeting Gram-negative and anaerobic early bacterial overgrowth and translocation. In a prospective observational study, the investigators recently suggested a protective effect of systematic oral antibiotics in terms of intestinal preservation, yielding a reduced occurrence of IN (HR: 0.16, 95% confidence interval 0.03-0.62). However, the systematic use of oral antibiotics in AMI remains controversial due to the individual and collective risk of increasing the carriage of multi-drug resistant bacterias.

DETAILED DESCRIPTION:
After the screening visit and informed consent collected by the recruiting investigator, all consecutive eligible patients (who will meet all inclusion criteria and none of exclusion criteria) will be included and randomized double-blind to oral antibiotics or double placebo group.

Patients will be evaluated at days 1, 3, 7, 14, 21 and 30 after the randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 and less 90
* AMI of arterial occlusive origin, defined by the combination of

  1. Onset < 7 days of clinical, biological and/or radiological signs of acute intestinal injury in the territory of at least superior mesenteric ischemia, including right-side colitis,
  2. significant vascular obstruction > 75% of the superior mesenteric artery, and
  3. no alternative diagnosis
* Admitted to the SURVI care network (Beaujon Hospital intensive care unit or SURVI, Bichat intensive care unit or vascular surgery department)

Exclusion Criteria:

* Other forms of mesenteric ischemia (chronic without acute manifestations, venous, non-occlusive, strangulation, aortic dissection)
* Isolated left-side ischemic colitis
* Mesenteric vascular lesion without small bowel injury or right colon
* Not eligible for vascular or digestive surgery or intensive care (palliative context)
* Indication for an emergency surgical intestinal resection at the admission to the SURVI care network
* Indication for urgent systemic antibiotic treatment on admission (evidence of sepsis defined as a SOFA score of 2 or more associated with an infection)
* Systemic or oral antibiotic therapy within 7 days before inclusion
* Known hypersensitivity to the active substance /excipients
* Contraindications to the investigational medicinal products (gentamicin, metronidazole)
* Unable to give consent (under guardianship or curatorship)
* Subject deprived of freedom, subject under a legal protective measure
* Patient refusal to participate
* Non-affiliation to a social security regimen or CMU
* Patient under State Medical Aid
* Pregnant or breastfeeding women
* Participation in another clinical study involving investigational medicinal product or patient being in the exclusion period at the end of a previous study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the efficacy of oral antibiotics compared to placebo on reducing the rate of intestinal necrosis or death (composite primary outcome) in AMI patients within 30 days following the randomisation. | 30 days after randomisation
  Occurrence of intestinal necrosis or death within 30 days following randomisation defined by the following criteria histology assessment OR all-cause mortality within 30 days following randomisation

SECONDARY OUTCOMES:
the rate of intestinal necrosis in the 30 days following the randomisation | 30 days after randomisation
  occurrence of intestinal necrosis within the 30 days following the randomisation.
the rate of short bowel syndrome (<200cm of remnant small bowel) at day-30 following the randomisation | 30 days after randomisation
  short bowel syndrome at day-30 after the randomisation
the length of intestinal resection at day-30 following the randomisation | 30 days after randomisation
  total length of intestinal resection at day 30 following the randomisation
the occurrence of organ failures within the 30 days following the randomisation | 30 days after randomisation
  occurrence of organ failure within the 30 days following the randomisation
the length of ICU stay | 30 days after randomisation
  number of days in the intensive care unit
the length of hospital stay | 30 days after randomisation
  number of hospitalization days
expected minor side effects during the 14 days of treatment | 14 days after randomisation
  Occurrence of minor side effects
hypersensitivity reactions during the 14 days of treatment | 14 days after randomisation
  Occurrence of hypersensitivity reaction to antibiotics
unexpected or serious adverse event throughout the duration of the study | 30 days after randomisation
  Occurrence of other adverse events
the occurrence of healthcare-associated infection | 30 days after randomisation
  Occurrence of healthcare-associated infection
the gentamicin during the 14 days of treatment | 14 days after randomisation
  Blood levels of gentamicin at randomisation day , days 7 and 14 after randomisation
the metronidazole during the 14 days of treatment | 14 days after randomisation
  Blood levels of metronidazole at randomisation day, days 7 and 14 after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Annabelle METOIS, Mrs, Study Chair — APHP
Locations (4):
- France (4):
  - Gastroentérologie-Hépatologie Beaujon, Clichy, France
  - Réanimation - Beaujon, Clichy, France
  - Chirurgie vasculaire, Paris, France
  - Réanimation Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: No